CLINICAL TRIAL: NCT00638326
Title: 150 mg Maintenance Dose of Clopidogrel in Patients With High On-Clopidogrel Platelet Reactivity After Elective Percutaneous Coronary Intervention
Brief Title: Doubling the Maintenance Dose of Clopidogrel in Patients With High On-Clopidogrel Platelet Reactivity
Acronym: DOSER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Greater differences between randomized patients than previously anticipated
Sponsor: University of Pecs (Other)
Responsible Party: Ivan G. Horvath, Heart Institute, University of Pécs, Dept. of Interventional Cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pecs-001
Record Dates: First submitted 2008-03-11; First posted 2008-03-19 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Stable Angina Pectoris; Ad Hoc Percutaneous Coronary Intervention
Keywords: Clopidogrel, thrombosis, Percutaneous Transluminal Coronary Angioplasty, stents
MeSH Terms: conditions — Angina, Stable; Thrombosis | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Patients who show adequate response to 600 mg loading dose of clopidogrel and receive standard 1x75 mg clopidogrel
- 2 (Experimental): Patients who show suboptimal response to 600 mg loading dose of clopidogrel and receive 1x150 mg clopidogrel for 28 days
  Interventions: Drug: clopidogrel
- 3 (Active Comparator): Patients who show suboptimal response to 600 mg loading dose of clopidogrel and receive 1x75 mg clopidogrel
  Interventions: Drug: clopidogrel plus placebo

INTERVENTIONS:
Drug: clopidogrel — 150 mg maintenance dose (2 capsules of 75 mg clopidogrel) for 28 days followed by standard 75 mg clopidogrel for one year
  Arms: 2
Drug: clopidogrel plus placebo — 75 mg maintenance dose (one capsule of 75 mg clopidogrel and one capsule placebo) for 28 days followed by standard 75 mg clopidogrel for one year
  Arms: 3

SUMMARY:
The purpose of the study is to determine whether administration of 150 mg clopidogrel is effective in reducing the one-year incidence of thromboischemic events in patients with high on-clopidogrel platelet reactivity compared to 75 mg clopidogrel after elective percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clopidogrel-naïve stable angina pectoris (CCS I-III)
* Coronary angiography that reveals significant DE NOVO coronary stenosis (diameter stenosis greater than 50% in two independent projections) feasible for ad hoc stent implantation

Exclusion Criteria:

* Acute coronary syndrome (STEMI, NSTEMI or unstable angina)
* Administration of clopidogrel/ticlopidine/coumarin in the past 6 weeks
* Contraindication to antiplatelet therapy
* Significant LM stenosis
* PCI due to instent restenosis
* Lesion located in bypass grafts
* Stroke in past one year
* Reduced life expectancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Cardiac death or non-fatal myocardial infarction or ischemia-driven target vessel revascularisation. | 12 months

SECONDARY OUTCOMES:
Academic Research Consortium (ARC) definite / probable stent thrombosis | 12 months
Cardiac death and non-fatal myocardial infarction | 12 months
Cardiac death or non-fatal myocardial infarction or ischemia-driven target vessel revascularisation or TIMI major/minor bleeding | 12 months
5 microM ADP-induced platelet aggregation assessed by light transmission aggregometer | 25 +/-2 days
VASP-PRI | 25 +/-2 days

CONTACTS AND LOCATIONS:
Overall Officials: Ivan G Horvath, MD PhD, Principal Investigator — Heart Institute, University of Pécs, HUNGARY; Daniel Aradi, MD, Study Director — Heart Institute, University of Pécs, HUNGARY; Andras Komocsi, MD PhD, Study Chair — Heart Institute, University of Pécs, HUNGARY
Locations (1):
- Heart Institute, University of Pécs, Dept. of Interventional Cardiology, Pécs, Hungary

REFERENCES:
- [Derived] Aradi D, Rideg O, Vorobcsuk A, Magyarlaki T, Magyari B, Konyi A, Pinter T, Horvath IG, Komocsi A. Justification of 150 mg clopidogrel in patients with high on-clopidogrel platelet reactivity. Eur J Clin Invest. 2012 Apr;42(4):384-92. doi: 10.1111/j.1365-2362.2011.02594.x. Epub 2011 Sep 9. PMID 21902692
- [Derived] Rideg O, Komocsi A, Magyarlaki T, Tokes-Fuzesi M, Miseta A, Kovacs GL, Aradi D. Impact of genetic variants on post-clopidogrel platelet reactivity in patients after elective percutaneous coronary intervention. Pharmacogenomics. 2011 Sep;12(9):1269-80. doi: 10.2217/pgs.11.73. Epub 2011 Aug 1. PMID 21806387